CLINICAL TRIAL: NCT04369222
Title: The Copenhagen Analgesic Study
Acronym: COPANA
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Anders Juul, Professor, Rigshospitalet, Denmark
Other Study IDs: COPANA5064
Record Dates: First submitted 2020-04-20; First posted 2020-04-30 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Gonad Regulating Hormone Adverse Reaction; Analgesic Adverse Reaction
MeSH Terms: interventions — Watchful Waiting; Acetaminophen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA EDTA-Blood Serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Controls: Children born from mothers with no consumption of mild analgesics 3 months before or during pregnancy
- Exposed: Children born from mothers with consumption of mild analgesics 3 months before or during pregnancy
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Maternal consumption of mild analgesics
  Other Names: Acetaminophen; Non steroidal antiinflammatory drugs; Acetyl salicylic acid
  Groups: Exposed

SUMMARY:
Fundamental aspects of reproductive function are established in fetal life and there is a present increased awareness of the potential effects of fetal exposures on reproductive health of offspring. Experimental studies strongly suggest detrimental effects of prenatal exposure to mild analgesics such as acetaminophen (e.g. paracetamol) and non-steroidal anti-inflammatory drugs, NSAIDs (e.g. ibuprofen and acetylsalicylic acid) on male as well as female gonadal development. Declining fertility has become a growing problem in developing countries, potentially resulting in severe socioeconomic challenges, and fetal exposure of mild analgesics causes part of these alarming observations.This is the first prospective human study designed primarily to assess the effect of fetal exposure of mild analgesics on male and female reproductive function.

DETAILED DESCRIPTION:
Fetal gonadal development is essential for adult reproductive health. Experimental studies strongly suggest that maternal use of mild analgesics (e.g. paracetamol and non-steroidal anti-inflammatory drugs (NSAIDs)) during pregnancy affect fetal gonadal development with possible severe reproductive repercussions.

In rodents, paracetamol and NSAIDs administered in therapeutic doses in early and mid-pregnancy are endocrine disruptive in the fetus causing reduced prostaglandin synthesis and delayed transition from germ cell mitosis to meiosis resulting in fetal germ cell apoptosis in both female and male gonads. Female offspring were born with reduced ovarian weight and concerning reduction (40-50%) in number of ovarian follicles. Females are born with a defined number of follicles that depletes throughout their reproductive lifespan, inevitably leading to menopause. Establishment of the primordial follicle pool during fetal life is therefore essential for female reproductive health and disruption of this process has important and lasting consequences. Although spermatogenesis is not restricted to fetal life, essential aspects of male gonadal development are tightly regulated in utero and in rodents exposure to mild analgesics causes decreased testosterone production and decreased fertility in male offspring.

In adulthood, exposed animals exhibited longer time to conceive and gave birth to fewer pubs per litter compared with controls. Furthermore, studies of rodents suggest that in both males and females, adverse reproductive effects are passed on to the next generation indicating altered genetic programming, i.e. epigenetic changes.

Analgesics are sold over the counter and up to 56% of pregnant women use mild analgesics during pregnancy. The bioavailability of acetaminophen is high (app. 90%), and the reactive metabolite passes freely over the placenta to the fetus.

Declining fertility has become a growing problem in developing countries, potentially resulting in severe socioeconomic challenges.

The anogenital distance (AGD) is defined as the distance from the anus to genital tubercle and is strongly affected by androgens in fetal life resulting in a longer AGD in males than in females.

The AGD has shown to be a sensitive marker of androgen exposure in fetal life, and remains the most sensitive parameter when evaluating prenatal exposure to endocrine disruptive environmental agents. Therefore, AGD has been identified as an endpoint in the US Environmental Protection Agency guidelines for reproductive toxicity studies.

In humans, use of mild analgesic during the first and second trimester was associated with reduced male AGD, congenital cryptorchidism and hypospadias suggestive of insufficient androgenic action. In male infants born with hypospadias, the reduction in AGD can be seen as early as in the third trimester where fetal AGD is below the fifth percentile compared to normative fetal AGD data. Thus, fetal AGD may assist in early detection of insufficient androgenic action and genital abnormalities.

In adult life, consequences can be impaired testosterone production, sub- and infertility as well as testis cancer.

Assessment of reproductive function in early life - minipuberty Minipuberty is a term used to describe the transient activation of the hypothalamic-pituitary-gonadal (HPG) axis during infancy in both boys and girls and is a window of opportunity for diagnosis of endocrine disorders as well as future reproductive function. Reproductive hormones exert effects on target tissue resulting in follicle maturation, growth of breast tissue and thickening of uterine endometrium (females) as well as testicular- and penile growth (males). The minipuberty is followed by a quiescent period during mid childhood until pubertal reactivation of the HPG axis at pubertal onset.

To date, no prospective human studies have assessed the effect of analgesic exposure on reproductive function. The few retrospective studies that are published are hampered by recall bias and/or lack of thorough reproductive evaluation, and no studies have in detail assessed human female reproductive function after the use of mild analgesics during pregnancy.

ELIGIBILITY:
Inclusion criteria:

Infants:

* Singleton pregnancies
* Term pregnancy (week 37+0 to 42+0)

Parents:

* Maternal and paternal Caucasian origin
* Maternal pre-pregnancy BMI between 18 and 35 kg/m2

Exclusion criteria:

Infants:

• Fetal malformations or chromosomal disorders

Parents:

* Serious maternal illness, including pre-existing maternal diabetes or thyroid gland diseases
* Gestational diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study is a population based prospective cohort study of 600 families (healthy pregnant mothers, biological fathers and their healthy male/female offspring.
  Pregnant women, meeting the inclusion criteria, and the fathers-to-be followed at the Department of Obstetrics, Rigshospitalet will be invited to participate.
  There are two groups of participants in this study:
  1. Healthy infants recruited specifically for this study
  2. The parents, i.e. the mother and father, of the healthy infants
  The two groups will include the following numbers (approximately) of participants:
  1. 600 healthy infants (based on expected son to daughter ratio of 105 to 100 in Denmark, we expect approximately equal distribution of boys and girl).
  2. 600 mothers and 600 fathers of healthy infants
Sampling Method: Non-Probability Sample
Enrollment: 685 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Ovarian volume (female infants) | 2.5 months old
  Ovarian volumen, measured by abdominal ultrasound
Ovarian follicle count (female infants) | 2.5 months old
  Ovarian follicle count, measured by abdominal ultrasound
Blood sample (female infants) | 2.5 months old
  Serum metabolites Anti Müllarian Hormone (AMH)
Testes volumen (male infants) | 2.5 months old
  Testes volumen, measured by ultrasound
Blood sample (male infants) | 2.5 months old
  Serum metabolites testosterone, free testosterone.

SECONDARY OUTCOMES:
Length (male and female infants) | 2.5 months old
  Length in cm
Weight (male and female infants) | 2.5 months old
  Weight in kilograms
Head circumference (male and female infants) | 2.5 months old
  Head circumference measured with a measurement tape, mm.
Abdominal circumference (male and female infants) | 2.5 months old
  Abdonimal circumference measured with a measurement tape, mm.
Height (fathers) | Gestational week 12
  Height in cm, by stadiometer (Holtain Ltd, Crymych, UK) with a precision of 0.1 cm
Weight (fathers) | Gestational week 12
  Weight in kilograms, by digital scale with a precision of 0.1 kg (SECA delta, model 707)
Biceps skinfold (father) | Gestational week 12
  Skinfold measured above the biceps, measured in mm (Harpenden skinfold Caliper, British Indicators Ltd, London, UK)
Triceps skinfold(father) | Gestational week 12
  Skinfold measured above the triceps, measured in mm (Harpenden skinfold Caliper, British Indicators Ltd, London, UK)
Flank skinfold (father) | Gestational week 12
  Skinfold measured at the flank, measured in mm (Harpenden skinfold Caliper, British Indicators Ltd, London, UK)
Scapula skinfold (father) | Gestational week 12
  Skinfold measured below the scapula all on the left side, measured in mm (Harpenden skinfold Caliper, British Indicators Ltd, London, UK)
Biceps skinfold (male and female infants) | 2.5 months old
  Skinfold measured above the biceps, measured in mm (Harpenden skinfold Caliper, British Indicators Ltd, London, UK)
Triceps skinfold (male and female infants) | 2.5 months old
  Skinfold measured above the triceps, measured in mm (Harpenden skinfold Caliper, British Indicators Ltd, London, UK)
Flank skinfold (male and female infants) | 2.5 months old
  Skinfold measured at the flank, measured in mm (Harpenden skinfold Caliper, British Indicators Ltd, London, UK)
Scapula skinfold (male and female infants) | 2.5 months old
  Skinfold measured below the scapula all on the left side, measured in mm (Harpenden skinfold Caliper, British Indicators Ltd, London, UK)
Asphyxia, adverse events (newborn) | Retrieved from patient files postpartum within 1 year of study completion
  Asphyxia (yes/no)
Meconium, adverse events (newborn) | Retrieved from patient files postpartum within 1 year of study completion
  Meconium in amionic fluids (yes/no)
Partus mode | Retrieved from patient files postpartum within 1 year of study completion
  Partus mode (vaginal delivery, cesarean section, instrumental delivery) (yes/no)
Birth weight (newborn) | Retrieved from patient files postpartum within 1 year of study completion
  Birth weight, grams
Birth length (newborn) | Retrieved from patient files postpartum within 1 year of study completion
  Birth length, cm
Gestational age (newborn) | Retrieved from patient files postpartum within 1 year of study completion
  Gestational age at birth, weeks and days
Drug intake (mother) | Retrieved from patient questionnaire postpartum within one year
  Pre- and perinatal drug intake, filled in by mother during the whole prengancy every two weeks online
Pregnancy outcome, preeclampsia (mother) | Retrieved from patient files postpartum within one year
  Preeclampsia (yes/no)
Pregnancy outcome, gestational hypertension (mother) | Retrieved from patient files postpartum within one year
  Gestational hypertension (yes/no)
Pregnancy outcome, induction of labor (mother) | Retrieved from patient files postpartum within one year
  In duction of labor (yes/no)
Medical history and exposure (parents) | Retrived from questionnaire within a half year
  General- and reproductive health, the pregnancy, own birth weight, lifestyle, drinking and smoking habits from questionnaire
Pubertal history (parents) | Retrived from questionnaire within a half year
  Pubertal history including age at menarche, pubertal timing with regard to peers, age at menopause of the mother of the parents etc. from questionnaire
Blood sample (mother) | Gestational week 12 and 2.5 months postpartum
  Blood samples will be drawn from an antecubital vein and will be measured for steroid hormone metabolites and metabolites of reproductive hormones.
  Testosterone, androstenedione, dehydroepiandrosterone (DHEA), dehydroepiandrosterone sulphate (DHEAS), Estradiol, Estrone, Progesterone, 17-hydroxyprogesterone: in-house mass-spectrometry; Turboflow (LC-MS/MS).
  Luteinizing hormone (LH), follicle stimulating hormone (FSH), Sex hormone Binding Globulin (SHBG): Time-resolved immuno- flouroimmunoassay; Delfia, Turko, Finland.
  Inhibin B: Specific enzyme-linked immunosorbent assay; Beckman Coulter GenII. Anti- Müllerian hormone (AMH): Specific enzyme immuno-metric assay; Immunotech Beckman Coulter.
  INSL3: Time-resolved immuno- flouroimmunoassay. IGF-I and IGFBP-3 will be analyzed using an immunoassay (iSYS, iDS).
Urine sample (mother) | Gestational week 12 and 2.5 months postpartum
  The urine sample will be collected in a cup and analyzed for:
  Steroid hormone metabolites using in-house mass-spectrometry; Turboflow (LC-MS/MS).
  Glycoprotein hormones, specifically FSH and LH, using immunoassays.
  Endocrine disrupting chemicals, specifically phthalates, phenols, perfluorinated compounds and parabens also using in-house mass-spectrometry; Turboflow (LC-MS/MS).
Blood sample (father) | Gestational week 12
  Blood samples will be drawn from an antecubital vein and will be measured for steroid hormone metabolites and metabolites of reproductive hormones:
  Testosterone, androstenedione, dehydroepiandrosterone (DHEA), dehydroepiandrosterone sulphate (DHEAS), Estradiol, Estrone, Progesterone, 17-hydroxyprogesterone: in-house mass-spectrometry; Turboflow (LC-MS/MS).
  Luteinizing hormone (LH), follicle stimulating hormone (FSH), Sex hormone Binding Globulin (SHBG): Time-resolved immuno- flouroimmunoassay; Delfia, Turko, Finland.
  Inhibin B: Specific enzyme-linked immunosorbent assay; Beckman Coulter GenII. Anti- Müllerian hormone (AMH): Specific enzyme immuno-metric assay; Immunotech Beckman Coulter.
  INSL3: Time-resolved immuno- flouroimmunoassay. IGF-I and IGFBP-3 will be analyzed using an immunoassay (iSYS, iDS).
Urine sample (father) | Gestational week 12
  The urine sample will be collected in a cup and analyzed for:
  Steroid hormone metabolites using in-house mass-spectrometry; Turboflow (LC-MS/MS).
  Glycoprotein hormones, specifically FSH and LH, using immunoassays.
  Endocrine disrupting chemicals, specifically phthalates, phenols, perfluorinated compounds and parabens also using in-house mass-spectrometry; Turboflow (LC-MS/MS).
Anogenital distance (AGD) (male and female infants) | 2.5 months old
  Distance from anus to genital tubercle, measured in mm with a ruler
Anogenital distance (AGD) (male and female infants) | App. gestational age 30 weeks
  Distance from anus to genital tubercle, third trimester ultrasound
Blood sample (female infants) | 2.5 months old
  (estradiol and inhibin B, luteinizing hormone (LH)/follicular stimulating hormone (FSH) ratio)
Blood sample (male infants) | 2.5 months old
  Serum metabolites of reproductive hormones (AMH, inhibin B levels, ratios of inhibin B/FSH and LH/FSH)
Classification of external genitalia with an external masculinization score (EMS) (male and female infants). EMS provides an objective aggregate score of the extent of masculinization of the external genitalia. | 2.5 months old
  It is an individual score with a maximum of 12 points. The following is assessed:
  Classification of genital tubercle, measured length with a ruler (mm) >30mm = 3 points, 21-30mm = 2 points, 11-20mm = 1 point,< 10mm = 0 points) Location of gonads, (objectively assessed): labioscrotal = 1,5 points, inguino-scrotal = 1, inguinal = 0,5 points, impalpable = 0 points Site of the urinary meatus (objectively assessed): typical male = 3 points, coronal/glandular = 2,5 points, penile = 2 points, peno-scrotal = 1,5 points, perineal = 0,5 points, typical female = 0 points.
  Labia/scrotal fusion (objectively assessed): fused = 3 points, posterior fusion = 1,5 points, unfused = 0 points.
Pubertal staging (male and female infants) | 2.5 months old
  Pubertal staging using Tanners classification (including testicular size in boys assessed by Prader's orchidometer)
Penile measurements (male infants) | 2.5 months old
  Penile measurements with a ruler
Epigenetic profiling (male and female infants) | Single determination, 2.5 months old
  Epigenetic variation of loci regulating hormone signalling
Urine sample (10 mL) (male and female infants) | 2.5 months old
  Steroid hormone metabolites using in-house mass-spectrometry; Turboflow (LC-MS/MS).
  Glycoprotein hormones, specifically FSH and LH, using immunoassays.
  Endocrine disrupting chemicals, specifically phthalates, phenols, perfluorinated compounds and parabens also using in-house mass-spectrometry; Turboflow (LC-MS/MS).
Medical report (mother) | Every 2 weeks from enrollment in early pregnancy to birth
  Specific medical report on medicine consumption incl. analgesics
Genetic profiling (male and female infants) | Single determination, 2.5 months old
  Genotyping of different genetic loci (genetic variation of loci regulating) hormone signalling, e.g. FSHB, etc.
Endometrial thickness (female infants) | 2.5 months old
  Endometrial thickness, measured by abdominal ultrasound
Uterine volume (female infants) | 2.5 months old
  Uterine volume, measured by abdominal ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Anders Juul, Professor, Principal Investigator — Department of Growth and Reproduction, Rigshospitalet
Locations (2):
- Denmark (2):
  - Department of Growth and Reproduction, Rigshospitalet, Copenhagen
  - Department of Obstetrics and Section of fetal medicine, Rigshospitalet, Copenhagen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dean A, van den Driesche S, Wang Y, McKinnell C, Macpherson S, Eddie SL, Kinnell H, Hurtado-Gonzalez P, Chambers TJ, Stevenson K, Wolfinger E, Hrabalkova L, Calarrao A, Bayne RA, Hagen CP, Mitchell RT, Anderson RA, Sharpe RM. Analgesic exposure in pregnant rats affects fetal germ cell development with inter-generational reproductive consequences. Sci Rep. 2016 Jan 27;6:19789. doi: 10.1038/srep19789. PMID 26813099
- [Background] Arendrup FS, Mazaud-Guittot S, Jegou B, Kristensen DM. EDC IMPACT: Is exposure during pregnancy to acetaminophen/paracetamol disrupting female reproductive development? Endocr Connect. 2018 Jan;7(1):149-158. doi: 10.1530/EC-17-0298. Epub 2018 Jan 5. PMID 29305399
- [Background] Kristensen DM, Mazaud-Guittot S, Gaudriault P, Lesne L, Serrano T, Main KM, Jegou B. Analgesic use - prevalence, biomonitoring and endocrine and reproductive effects. Nat Rev Endocrinol. 2016 Jul;12(7):381-93. doi: 10.1038/nrendo.2016.55. Epub 2016 May 6. PMID 27150289
- [Background] Kristensen DM, Hass U, Lesne L, Lottrup G, Jacobsen PR, Desdoits-Lethimonier C, Boberg J, Petersen JH, Toppari J, Jensen TK, Brunak S, Skakkebaek NE, Nellemann C, Main KM, Jegou B, Leffers H. Intrauterine exposure to mild analgesics is a risk factor for development of male reproductive disorders in human and rat. Hum Reprod. 2011 Jan;26(1):235-44. doi: 10.1093/humrep/deq323. Epub 2010 Nov 8. PMID 21059752
- [Background] Holm JB, Mazaud-Guittot S, Danneskiold-Samsoe NB, Chalmey C, Jensen B, Norregard MM, Hansen CH, Styrishave B, Svingen T, Vinggaard AM, Koch HM, Bowles J, Koopman P, Jegou B, Kristiansen K, Kristensen DM. Intrauterine Exposure to Paracetamol and Aniline Impairs Female Reproductive Development by Reducing Follicle Reserves and Fertility. Toxicol Sci. 2016 Mar;150(1):178-89. doi: 10.1093/toxsci/kfv332. Epub 2016 Jan 5. PMID 26732887
- [Background] BAKER TG. A QUANTITATIVE AND CYTOLOGICAL STUDY OF GERM CELLS IN HUMAN OVARIES. Proc R Soc Lond B Biol Sci. 1963 Oct 22;158:417-33. doi: 10.1098/rspb.1963.0055. No abstract available. PMID 14070052
- [Background] Reel JR, Lawton AD, Lamb JC 4th. Reproductive toxicity evaluation of acetaminophen in Swiss CD-1 mice using a continuous breeding protocol. Fundam Appl Toxicol. 1992 Feb;18(2):233-9. doi: 10.1016/0272-0590(92)90051-i. PMID 1601223
- [Background] Johansson HK, Jacobsen PR, Hass U, Svingen T, Vinggaard AM, Isling LK, Axelstad M, Christiansen S, Boberg J. Perinatal exposure to mixtures of endocrine disrupting chemicals reduces female rat follicle reserves and accelerates reproductive aging. Reprod Toxicol. 2016 Jun;61:186-94. doi: 10.1016/j.reprotox.2016.03.045. Epub 2016 Apr 2. PMID 27049580
- [Background] Ersboll AS, Hedegaard M, Damm P, Johansen M, Tabor A, Hegaard HK. Changes in the pattern of paracetamol use in the periconception period in a Danish cohort. Acta Obstet Gynecol Scand. 2015 Aug;94(8):898-903. doi: 10.1111/aogs.12667. Epub 2015 May 29. PMID 25939806
- [Background] Lind DV, Main KM, Kyhl HB, Kristensen DM, Toppari J, Andersen HR, Andersen MS, Skakkebaek NE, Jensen TK. Maternal use of mild analgesics during pregnancy associated with reduced anogenital distance in sons: a cohort study of 1027 mother-child pairs. Hum Reprod. 2017 Jan;32(1):223-231. doi: 10.1093/humrep/dew285. Epub 2016 Nov 16. PMID 27852690
- [Background] Rebordosa C, Zelop CM, Kogevinas M, Sorensen HT, Olsen J. Use of acetaminophen during pregnancy and risk of preeclampsia, hypertensive and vascular disorders: a birth cohort study. J Matern Fetal Neonatal Med. 2010 May;23(5):371-8. doi: 10.3109/14767050903334877. PMID 19929241
- [Background] Nitsche JF, Patil AS, Langman LJ, Penn HJ, Derleth D, Watson WJ, Brost BC. Transplacental Passage of Acetaminophen in Term Pregnancy. Am J Perinatol. 2017 May;34(6):541-543. doi: 10.1055/s-0036-1593845. Epub 2016 Nov 2. PMID 27806383
- [Background] Myrskyla M, Kohler HP, Billari FC. Advances in development reverse fertility declines. Nature. 2009 Aug 6;460(7256):741-3. doi: 10.1038/nature08230. PMID 19661915
- [Background] Tromp M, Ravelli AC, Reitsma JB, Bonsel GJ, Mol BW. Increasing maternal age at first pregnancy planning: health outcomes and associated costs. J Epidemiol Community Health. 2011 Dec;65(12):1083-90. doi: 10.1136/jech.2009.095422. Epub 2010 Aug 13. PMID 20709858
- [Background] Gallavan RH Jr, Holson JF, Stump DG, Knapp JF, Reynolds VL. Interpreting the toxicologic significance of alterations in anogenital distance: potential for confounding effects of progeny body weights. Reprod Toxicol. 1999 Sep-Oct;13(5):383-90. doi: 10.1016/s0890-6238(99)00036-2. PMID 10560587
- [Background] Juul A, Almstrup K, Andersson AM, Jensen TK, Jorgensen N, Main KM, Rajpert-De Meyts E, Toppari J, Skakkebaek NE. Possible fetal determinants of male infertility. Nat Rev Endocrinol. 2014 Sep;10(9):553-62. doi: 10.1038/nrendo.2014.97. Epub 2014 Jun 17. PMID 24935122
- [Background] Dean A, Sharpe RM. Clinical review: Anogenital distance or digit length ratio as measures of fetal androgen exposure: relationship to male reproductive development and its disorders. J Clin Endocrinol Metab. 2013 Jun;98(6):2230-8. doi: 10.1210/jc.2012-4057. Epub 2013 Apr 8. PMID 23569219
- [Background] Leverrier-Penna S, Mitchell RT, Becker E, Lecante L, Ben Maamar M, Homer N, Lavoue V, Kristensen DM, Dejucq-Rainsford N, Jegou B, Mazaud-Guittot S. Ibuprofen is deleterious for the development of first trimester human fetal ovary ex vivo. Hum Reprod. 2018 Mar 1;33(3):482-493. doi: 10.1093/humrep/dex383. PMID 29408962
- [Background] Snijder CA, Kortenkamp A, Steegers EA, Jaddoe VW, Hofman A, Hass U, Burdorf A. Intrauterine exposure to mild analgesics during pregnancy and the occurrence of cryptorchidism and hypospadia in the offspring: the Generation R Study. Hum Reprod. 2012 Apr;27(4):1191-201. doi: 10.1093/humrep/der474. Epub 2012 Feb 2. PMID 22301570
- [Background] Gilboa Y, Perlman S, Kivilevitch Z, Messing B, Achiron R. Prenatal Anogenital Distance Is Shorter in Fetuses With Hypospadias. J Ultrasound Med. 2017 Jan;36(1):175-182. doi: 10.7863/ultra.16.01006. Epub 2016 Nov 28. PMID 27925677
- [Background] Mendiola J, Stahlhut RW, Jorgensen N, Liu F, Swan SH. Shorter anogenital distance predicts poorer semen quality in young men in Rochester, New York. Environ Health Perspect. 2011 Jul;119(7):958-63. doi: 10.1289/ehp.1103421. Epub 2011 Mar 4. PMID 21377950
- [Background] Kuiri-Hanninen T, Sankilampi U, Dunkel L. Activation of the hypothalamic-pituitary-gonadal axis in infancy: minipuberty. Horm Res Paediatr. 2014;82(2):73-80. doi: 10.1159/000362414. Epub 2014 Jul 5. PMID 25012863
- [Background] Lanciotti L, Cofini M, Leonardi A, Penta L, Esposito S. Up-To-Date Review About Minipuberty and Overview on Hypothalamic-Pituitary-Gonadal Axis Activation in Fetal and Neonatal Life. Front Endocrinol (Lausanne). 2018 Jul 23;9:410. doi: 10.3389/fendo.2018.00410. eCollection 2018. PMID 30093882
- [Derived] Fischer MB, Mola G, Rom AL, Frederiksen H, Johannsen TH, Sundberg K, Hegaard HK, Juul A, Hagen CP. Ovarian and Uterine Morphology in Minipuberty: Associations With Reproductive Hormones: a COPANA Study of 302 Girls. J Clin Endocrinol Metab. 2025 Mar 17;110(4):1015-1022. doi: 10.1210/clinem/dgae678. PMID 39329336